CLINICAL TRIAL: NCT03575143
Title: Obstructive Sleep Apnea Endotypes and Impact on Phenotypes of People Living With HIV
Acronym: PLWH/OSA
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert L. Owens, Associate Clinical Professor, University of California, San Diego
Other Study IDs: 180160; R01HL142114 (NIH)
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Human Immunodeficiency Virus; Obstructive Sleep Apnea
Keywords: HIV; OSA; PLWH; Sleep; Obstructive Sleep Apnea; Human Immunodeficiency Virus; CPAP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Approximately 10-15 cc of blood will be drawn in the morning at wake into serum separator and EDTA tubes. Serum samples will be immediately processed to separate serum, which will be stored in darkness at -70 F to preserve until analysis can be conducted. EDTA tubes will be processed and refrigerated for use within 24 hours. Blood will also be collected to measure high sensitivity C Reactive Protein (hsCRP), insulin, glucose (to calculate HOMA-IR), cytokines such as IL-6 and TNF-alpha.119 The investigators will also store plasma for other potential markers, to explore other interactions, such as markers of liver disease like ALT and AST.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PLWH+OSA: Subjects diagnosed with both Human Immunodeficiency Virus and Obstructive Sleep Apnea based on overnight sleep study
- PLWH-OSA: Subjects diagnosed with both Human Immunodeficiency Virus without Obstructive Sleep Apnea based on overnight sleep study
- PLWH?OSA: Those who signed consent but did not complete all the baseline assessments and overnight sleep study

SUMMARY:
The investigators seek to understand how the different underlying causes of OSA affect the way people living with HIV (PLWH) experience OSA. The investigators also want to understand how symptoms of obstructive sleep apnea improve with treatment, and if this too, is affected by the underlying cause of OSA in that individual

DETAILED DESCRIPTION:
Overnight Visit #1. Subjects will arrive to the research sleep laboratory at approximately 7PM and undergo the following procedures:

1. Polysomnography: Monitoring for standard clinical polysomnography study will be applied to the subject, as follows: The subject will have EEG, EMG, EOG, and ECG electrodes, an adhesive body position sensor placed in standard locations. Pulse oximetry sensor will be attached either to a finger or ear lobe and secured by tape. The following parameters will be measured during sleep: electroencephalogram, eye movement, electrocardiogram, electromyogram, leg movement, snoring sounds, nasal pressure, and nasal-oral airflow by thermistor, respiratory effort and body position by piezo-electric bands of the thorax and abdomen or magnetometers, position sensors, and pulse oximetry. This equipment is standard for diagnostic polysomnography and should not be uncomfortable.

   Once all of this equipment has been comfortably and securely fastened, the subject will be allowed to fall asleep and data recording will begin. Subjects will be asked to remain in the supine position as much as possible. All data will be acquired on a 1401 plus interface and Spike 2 software. The study will end at approximately 6 AM, at which time the monitoring equipment will be removed, and the subject will undergo a blood draw in this fasting state.
2. Phlebotomy: Venipuncture will be performed by a certified research staff or physician using standard techniques and appropriate blood borne pathogen precautions. Approximately 10-15 cc of blood will be drawn in the morning at wake into serum separator and EDTA tubes. Serum samples will be immediately processed to separate serum, which will be stored in darkness at -70 F to preserve until analysis can be conducted. EDTA tubes will be processed and refrigerated for use within 24 hours. Blood will also be collected to measure high sensitivity C Reactive Protein (hsCRP), insulin, glucose (to calculate HOMA-IR), cytokines such as IL-6 and TNF-alpha.119 The investigators will also store plasma for other potential markers, to explore other interactions, such as markers of liver disease like ALT and AST.

Subjects will then be able to go home. They will leave the actiwatch for the investigators. The investigators anticipate that Overnight Visit #1 will last 10 hours (most of which will be spent asleep).

If subjects are not found to have OSA, they will not continue with the study. (End of Aim #1)

Aims #2 and #3 Subjects found to have OSA (with AHI >5 events/hour) will be referred for clinical evaluation (by a sleep physician not involved in the study) and treatment, and will also return for overnight visit #2, and continue to be followed with weekly phone calls and a repeat assessment 3 months after starting OSA treatment.

Overnight Visit #2 (Aim #2) Measurement of Endotypic Traits

This visit will be scheduled to occur within 1 month of visit 1, and will be prior to any clinical OSA treatment. Subjects will come to the sleep research laboratory about 2-3 hours before their usual bedtime. They will undergo polysomnography, as described above, without the physiological CPAP testing procedure. To review, the subject will have EEG, EMG, EOG, and ECG electrodes, an adhesive body position sensor placed in standard locations. Pulse oximetry sensor will be attached either to a finger or ear lobe and secured by tape. The following parameters will be measured during sleep: electroencephalogram, eye movement, electrocardiogram, electromyogram, leg movement, snoring sounds, nasal pressure, and nasal-oral air flow by thermistor, respiratory effort and body position by piezo-electric bands of the thorax and abdomen or magnetometers, position sensors, and pulse oximetry. This equipment is standard for diagnostic polysomnography and should not be uncomfortable.

Additional equipment for the physiological sleep study will also be applied to the subject, as follows:

A thin esophageal catheter (6-8 french) with an electrode array to measure diaphragm electromyography will be placed via the nares. Prior to the cannula placement the subject will received 2 sprays of a nasal decongestant (0.05% oxymetazoline hydrochloride), followed by 4% lidocaine topical spray for local anesthesia. The catheter will be confirmed to be in the proper position by examining the signal, then taped to the nose (and later secured to the CPAP mask). The esophageal catheter placement may be omitted by subject or investigator request; in this case subjects can still remain in the study.

A standard CPAP mask will be placed over the nose and secured with velcro straps. If necessary, the subject's mouth will be either taped closed or a chin strap applied to ensure nasal breathing. A specially modified continuous positive airway pressure (CPAP) device (ResMed, San Diego, CA) that delivers both positive and negative airway pressure will be connected to the mask. Once all of this equipment has been comfortably and securely fastened, the subject will be allowed to fall asleep and data recording will begin. Subjects will be asked to remain in the supine position as much as possible. All data will be acquired on a 1401 plus interface and Spike 2 software (Cambridge Electronics Design Ltd, Cambridge, UK).

After sleep onset, airway pressure will be increased in order to abolish flow limitation. During sleep, a previously validated sequence of pressure reductions will be performed in order to measure respiratory control and upper airway characteristics, as follows: The holding pressure will be abruptly changed to atmospheric pressure for several breaths, then returned to holding pressure. After a short time, the pressure will be gradually reduced over the course of several minutes, until an arousal occurs on the EEG (generally not associated with any awareness by the subject). The subject will be given several minutes to resume normal sleep, and the procedure will be repeated until three stable readings are obtained. Subsequently, the procedure will be repeated, but with a reduction in pressure to a level that does not induce arousal. After a short period of time with stable breathing at this pressure, the pressure will be returned to the holding pressure to measure ventilatory response. This will be repeated until 3 stable values are obtained.

The study will end at approximately 4 AM, at which time the monitoring equipment will be removed, and the subject will be allowed to go home. However, if the subject is still sleepy, they will be allowed to sleep with CPAP applied until they feel rested.

Aim #3 investigates the impact of CPAP on the phenotypic traits.

The investigators anticipate that Overnight Visit #2 will last 8 hours (most of which will be spent sleeping).

Weekly Phone calls: Subjects will be referred to a sleep physician for PAP therapy. The treatment is expected every day to be worn when participants are asleep (including naps). In addition to usual clinical care provided to ensure optimal adherence to PAP therapy, the research staff will be in weekly contact with subjects to provide encouragement, and identify and troubleshoot impediments to all-night, every-night use of PAP therapy. These phone calls will be 10-15 minutes each for 12 weeks.

2 weeks prior to returning for Daytime Visit #2, subjects will be mailed or delivered an actiwatch to wear for 2 weeks.

Daytime Visit #2: Impact of OSA treatment on Sleep and Activity Phenotypes

After three months of OSA treatment, subjects will return to the sleep lab to repeat all of the same measurements described under Visit 1 with the exception of the lung function testing (see Daytime Visit #1). This visit will generally occur in the morning at which time another fasting blood sample will be collected.

Additionally for subjects using PAP therapy for treatment of OSA, the investigators will obtain a PAP download which will report therapeutic holding pressure, residual apnea-hypopnea index, as well as multiple parameters of adherence such as days of use, number of days >4 hours per night, etc. Mask type (nasal vs. oronasal, etc) will be recorded. The actiwatch will be returned to the investigators to assess the impact of PAP therapy on activity levels, pattern of activity and sleep duration.

The investigators anticipate that Daytime Visit #2 will be 2 hours.

The total duration of the participant's involvement in the study is expected to be a total of 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of HIV and viral suppression
* Ages 18-65 years old
* BMI 20 - 35 kg/m2

Exclusion Criteria:

* Pregnancy
* Inability to complete study procedures, such as questionnaires that are only available/validated in English.
* Known OSA already on effective therapy and adherent to treatment
* Other known untreated sleep fragmenting disorder, such as periodic limb movement disorder, or narcolepsy. We will NOT exclude based on insomnia, given that OSA and insomnia frequently exist together.
* Chronic lung disease requiring the use of supplemental oxygen, or with evidence of hypercapnia due to obstructive lung disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with HIV on ART and demonstrated viral suppression will be recruited into the study to undergo a standard sleep study, a research sleep study, and other procedures designed to measure phenotypic expression of sleep/OSA. All of the planned experiments will take place at UCSD.
  This study does not contain any exclusion by race, gender or ethnicity. We will only study subjects able to give self-consent. Thus, patients with existing severe dementia, children, prisoners, etc. will not be included. We believe that duration of HIV infection, HIV medication use and duration of use may be potentially important. However, while we will gather such information as completely as possible, we will not limit participation based on these factors. Finally, our preliminary data suggest that many PLWH use medications that might affect sleep, such as benzodiazepines, cannabinoids, etc. We plan to INCLUDE these subjects to increase the generalizability of our findings.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Owens, MD, Principal Investigator — UCSD Pulmonary and Sleep Medicine
Locations (1):
- Altman Clinical and Translational Research Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berry DL, Orr JE, Schmickl CN, DeYoung P, Bosompra NO, Ancoli-Israel S, Grant I, Young-Karris M, Malhotra A, Owens RL. Effects of Treating Obstructive Sleep Apnea on Common Symptoms of HIV. J Acquir Immune Defic Syndr. 2025 Dec 15;100(5):454-461. doi: 10.1097/QAI.0000000000003753. PMID 40856602
- [Derived] Orr JE, Velazquez J, Schmickl CN, Bosompra NO, DeYoung PN, Gilbertson D, Malhotra A, Grant I, Ancoli-Israel S, Karris MY, Owens RL. Sleep, Sleep Apnea, and Fatigue in People Living With HIV. J Acquir Immune Defic Syndr. 2024 Oct 1;97(2):192-201. doi: 10.1097/QAI.0000000000003481. PMID 39250653
- [Derived] Schmickl CN, Bosompra NO, DeYoung PN, Gilbertson D, Orr JE, Malhotra A, Grant I, Ancoli-Israel S, Young MK, Owens RL. Diagnostic performance of screening tools for the detection of obstructive sleep apnea in people living with HIV. J Clin Sleep Med. 2022 Jul 1;18(7):1797-1804. doi: 10.5664/jcsm.9964. PMID 35383569

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects living with HIV were enrolled after written informed consent was obtained. Enrolled subjects completed daytime questionnaires, 1 week of actigraphy, and then an overnight sleep study. Enrolled subjects were placed into 3 different groups: 1) those with OSA (based on Medicare Criteria 4%)(PLWH+OSA), 2) those without OSA (PLWH-OSA), and 3) those who did not complete overnight testing (PLWH?OSA).
Groups:
- PLWH+OSA: Subjects diagnosed with both Human Immunodeficiency Virus and Obstructive Sleep Apnea
- PLWH-OSA: Subjects diagnosed with both Human Immunodeficiency Virus without Obstructive Sleep Apnea
Period: Overall Study
Arm/Group | PLWH+OSA | PLWH-OSA | PLWH?OSA
Started | 66 | 55 | 11
Completed | 66 | 55 | 0
Not Completed | 0 | 0 | 11
Not completed — Lost to Follow-up | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 5
Not completed — new information provide after consent, no longer met inclusion criteria | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- PLWH?OSA: Subjects diagnosed with HIV who signed consent but did not complete overnight sleep study
- Total: Total of all reporting groups
Arm/Group | PLWH+OSA | PLWH-OSA | PLWH?OSA | Total
Number analyzed (Participants) | 66 | 55 | 11 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 66 | 55 | 11 | 132
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 15 | 2 | 20
  Male | 63 | 40 | 9 | 112
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 0 | 5
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 10 | 9 | 3 | 22
  White | 44 | 32 | 6 | 82
  More than one race | 6 | 10 | 2 | 18
  Unknown or Not Reported | 2 | 1 | 0 | 3
Apnea Hypopnea Index (4%) [Mean (Standard Deviation); unit: events/hr] — The apnea hypopnea index is the total number of apneas and hypopneas measured during the overnight sleep study, divided by the total sleep time.
  Apneas refer to a complete cessation of airflow for at least 10 seconds.
  Hypopneas refer to reductions in airflow from baseline that lead to a reduction in oxygen saturation or arousal. Two commonly used definitions of hypopnea are:
  * hypopnea 4% - a greater than 30% decrease in nasal pressure accompanied by a 4% desaturation
  * hypopnea 3% - a greater than 30% decrement in nasal pressure with a 3% desaturation and/or an arousal from sleep Population: Subjects in the PLWH?OSA arm did not complete the baseline polysomnogram used to measure the apnea hypopnea index (3 or 4%).
  events/hr
    number analyzed (Participants) | 66 | 55 | 0 | 121
    (all) | 32 (23) | 2 (2) |  | 19 (23)
Apnea Hypopnea Index (3%) [Mean (Standard Deviation); unit: events/hr] — The apnea hypopnea index is the total number of apneas and hypopneas measured during the overnight sleep study, divided by the total sleep time.
  Apneas refer to a complete cessation of airflow for at least 10 seconds.
  Hypopneas refer to reductions in airflow from baseline that lead to a reduction in oxygen saturation or arousal. Two commonly used definitions of hypopnea are:
  * hypopnea 4% - a greater than 30% decrease in nasal pressure accompanied by a 4% desaturation
  * hypopnea 3% - a greater than 30% decrement in nasal pressure with a 3% desaturation and/or an arousal from sleep Population: Subjects in the PLWH?OSA arm did not complete the baseline polysomnogram used to measure the apnea hypopnea index (3 or 4%).
  events/hr
    number analyzed (Participants) | 66 | 55 | 0 | 121
    (all) | 42 (24) | 7 (6) |  | 26 (25)

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time Measured Using the Psychomotor Vigilance Task
Description: The Psychomotor Vigilance Task (PVT) is commonly used to asses the impact of sleep (or sleep deprivation) on cognitive performance. Subjects are instructed to respond (by tapping a key on a keyboard) as fast as possible to a graphical stimulus displayed on a computer screen. The stimulus is presented multiple times at variable intervals every few seconds for 10 minutes. The reaction time is the mean latency from appearance of the stimulus to the response by the participant. Higher values suggest a slower reaction time compared to lower values.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: ms
Groups:
- PLWH+OSA+High AT: Subjects diagnosed with both Human Immunodeficiency Virus and Obstructive Sleep Apnea with a High arousal threshold
- PLWH+OSA+Low AT: Subjects diagnosed with both Human Immunodeficiency Virus and Obstructive Sleep Apnea with a Low Arousal Threshold
- PLWH-OSA: Subjects diagnosed with Human Immunodeficiency Virus without Obstructive Sleep Apnea
Arm/Group | PLWH+OSA+High AT | PLWH+OSA+Low AT | PLWH-OSA
Number analyzed (Participants) | 35 | 24 | 51
ms | 346 (38) | 353 (39) | 348 (48)

2. Secondary Outcome: Reactive Hyperemia Index (RHI) Assessed by Peripheral Arterial Tonometry
Description: Reactive hyperemia is measured using the commercially available EndoPAT device (Itamar Medical). Briefly, the device uses finger plethysmography to measure the finger arterial pulse wave amplitude. Subjects have the pulse wave measured during rest, during the application of a blood pressure cuff to occlude blood flow for 5 minutes, and then once the blood pressure cuff is deflated. The reactive hyperemia index (RHI) is the ratio (thus dimensionless) of the pulse wave amplitude after occlusion compared to the pre-occlusion value. Values for the RHI are physiologically greater than 1 (least health endothelial function), with the highest values in the literature about 3. (See Itzhaki SLEEP 2005;28(5):594-600.) Higher ratios are considered to reflect healthier endothelial function.
Time Frame: 1 day
Population: A loop gain of .7 was used as a cutoff between Low and High LG groups
Measure: Mean (Standard Deviation); unit: ratio (unitless)
Groups:
- PLWH+OSA+Low LG: People diagnosed with Human Immunodeficiency Virus and Obstructive Sleep Apnea who have a Low Loop Gain (more stable ventilatory drive)
- PLWH+OSA+High LG: People diagnosed with Human Immunodeficiency Virus and Obstructive Sleep Apnea who have a High Loop Gain (less stable ventilatory drive)
Arm/Group | PLWH+OSA+Low LG | PLWH+OSA+High LG
Number analyzed (Participants) | 37 | 22
ratio (unitless) | 1.6 (.38) | 1.52 (.36)

3. Other Pre Specified Outcome: Neurocognitive and Endothelial Function After CPAP
Description: To test in PLWH+OSA whether 3 months of PAP treatment results in changes in OSA manifestations. This aim will allow us to test the hypothesis that endotype underlying OSA will be predictive of the specific clinical improvements seen in adherent users of PAP therapy. For example, those with high LG at baseline will have the greatest improvement in endothelial dysfunction with PAP therapy compared to other OSA patients with similar disease severity as measured by AHI.
Time Frame: 3 months
Reporting Status: Not Posted, anticipated posting 2023-12

ADVERSE EVENTS:
Time Frame: Duration of participation in the study, which varied according to each study participant. Those subjects who were PLWH-OSA completed the study generally in 7-10 days. Subjects who were PLWH+OSA completed an additional overnight sleep study and then used CPAP therapy for 12 weeks. Their participation in the study might be up to 6 months depending on the timing of procedures.
Arm/Group | PLWH+OSA | PLWH-OSA | PLWH?OSA
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/55 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/55 | 0/11
Other Adverse Events (participants affected / at risk) | 1/66 | 0/55 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLWH+OSA (N=66) | PLWH-OSA (N=55) | PLWH?OSA (N=11)
Epistaxis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — The subject reported epistaxis after starting CPAP.

LIMITATIONS AND CAVEATS:
Research and clinical procedures were interrupted by the COVID pandemic. In particular, the planned treatment phase (e.g. CPAP) of the study had greater than expected participant drop out and lower than expected adherence to CPAP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT03575143/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT03575143/SAP_001.pdf
  • Informed Consent Form (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT03575143/ICF_002.pdf